CLINICAL TRIAL: NCT07217301
Title: A Randomized, Open-Label, Multicenter, Phase 3 Study Evaluating the Efficacy and Safety of IBI363 Versus Docetaxel in Participants With Unresectable Locally Advanced or Metastatic Squamous Non-Small Cell Lung Cancer With Disease Progression on or After Platinum-Based Chemotherapy and Anti-PD-1/PD-L1 Immunotherapy
Brief Title: IBI363 vs Docetaxel in Patients With Advanced Squamous Lung Cancer After Standard Treatments Have Failed
Acronym: MarsLight-11
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fortvita Biologics (USA)Inc. (Industry)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363C301
Record Dates: First submitted 2025-08-31; First posted 2025-10-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: iO Resistant sqNSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IBI363 (Experimental): IBI363 is a first-in-class bispecific monoclonal antibody (mAb) comprised of an interleukin-2 (IL-2) mutein fused with a recombinant anti-programmed cell death protein 1 (anti-PD-1) mAb. IBI363 was precisely designed and constructed to afford targeted binding of tumor-specific CD8+ T cells (TSTs) that co-express PD-1 and CD25 (IL2Ra) receptors. The mechanism of action of IBI363 is blocking the PD-(L)1 and activating the IL-2 pathways simultaneously to reverse T cell exhaustion and promote activation of T cells and natural killer (NK) cells, and consequently eliminate tumor cells.
  Interventions: Drug: IBI363
- Control (Active Comparator): Docetaxel or comparable generic brand
  Interventions: Drug: Control Arm

INTERVENTIONS:
Drug: IBI363 — Investigational product will be administered by IV infusion
  Arms: IBI363
Drug: Control Arm — Comparator product will be administered by IV infusion
  Arms: Control

SUMMARY:
Phase: 3 Type: Randomized, open-label, multi-regional, multi-center Population: Adults with advanced/metastatic squamous Non Small Cell Lung Cancer (NSCLC), post-progression on platinum chemo + PD-1/PD-L1 immunotherapy Enrollment: ~600 participants Randomization: 1:1 (IBI363 vs. docetaxel)

Stratification factors:

1. Primary vs. acquired IO resistance
2. Concurrent vs. sequential prior chemo-immunotherapy
3. Region (Asia vs. non-Asia)

Treatment Arms:

1. IBI363 Arm (Investigational Drug):

   Priming dose: 0.1 mg/kg on Day 1 of Cycle 1 (C1D1) Intended dose: 3 mg/kg every 3 weeks (Q3W) starting Day 8 of Cycle 1 (C1D8) Cycle duration: 28 days for Cycle 1, then 21 days from Cycle 2 onward Dose adjustments: Up to 2 reductions (1.5 mg/kg or 1 mg/kg Q3W) allowed for adverse events (AEs) Re-priming protocol: Required if delays in dosing exceed defined thresholds (e.g., >10 days post-priming or ≥5 weeks since last dose)
2. Control Arm (Docetaxel):

75 mg/m² every 3 weeks (Q3W), starting from C1D1 21-day cycle duration Dose Reduction: as per label

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the written informed consent form and be able to comply with the visit schedule and related procedures specified in the protocol.
2. Male or female participants must be at least 18 years old or the legal age of majority in their country, whichever is greater.
3. Have locally unresectable advanced or metastatic histologically or cytologically confirmed squamous NSCLC Note: Mixed small cell carcinoma, or other pathological components are excluded.
4. Resistant or refractory to systemic anti-tumor therapy, including platinum-based doublet chemotherapy and primary or secondary resistance to anti-PD-1/PD-L1 monoclonal antibody given in combination or sequentially; or given as neoadjuvant and/or adjuvant therapy, which will be considered first-line treatment if the disease has recurred or progressed during such treatment or within 6 months after discontinuation.
5. Radiographic progression per RECIST v1.1 during or within 6 months after discontinuation of anti-PD-1/PD-L1 monoclonal antibody treatment.
6. Agree to provide archival (collected within 2 years before signing the informed consent form if biopsy cannot be performed or participant refuses fresh biopsy) tumor tissue specimens for PD-L1 expression level testing and exploratory analysis of other biomarkers.
7. Have at least one measurable lesion (target lesion) by computed tomography (CT) or magnetic resonance imaging (MRI) according to RECIST v1.1. Lesions that have previously received radiotherapy or intratumoral injection can be used as measurable lesions if they show progression after treatment (either tissue confirmed or more than 3 months after treatment) as per RECIST v1.1.
8. ECOG PS score of 0 or 1.
9. Expected survival time ≥ 3 months.
10. Women of childbearing potential (WOCBP) or men with female partners of childbearing potential must agree to take effective contraceptive measures during the entire course of treatment and for 6 months after the last dose of study treatment.
11. Lactating women must agree to strictly abstain from breastfeeding during the entire Treatment Period and for 6 months after the treatment.

Exclusion Criteria:

1. Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of any study drug. WOCBP or fertile men with WOCBP partner(s), not using and/or not willing to use a highly effective method of contraception.
2. Known actionable genomic alteration, including any of the following driver gene mutations:

   * Epidermal growth factor receptor (EGFR): including exon 19 deletion, exon 21 L858R, exon 20 T790M, exon 20 S768I, exon 21 L861Q, exon 18 G719X, and exon 20 insertion mutations.
   * Kirsten rate sarcoma virus (KRAS) G12C mutation.
   * Anaplastic lymphoma kinase (ALK) rearrangement.
   * ROS proto-oncogene 1, receptor tyrosine kinase (ROS1) rearrangement.
   * B-Raf proto-oncogene, serine/threonine kinase (BRAF) V600E mutation.
   * Neurotrophic tyrosine receptor kinase (NTRK) 1/2/3 fusion.
   * MET proto-oncogene, receptor tyrosine kinase (MET) exon 14 skipping mutation.
   * RET proto-oncogene (RET) rearrangement.
   * V-erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 (ERBB2, also known as HER2) mutation.
   * Other gene mutation types where a targeted therapy has been completely approved for marketing by a local regulatory authority.

   Note: It is not mandatory to have undergone driver gene testing.
3. Active or symptomatic brain metastases. Participants who are clinically and radiologically stable at least 4 weeks after treatment and participants with small, asymptomatic, incidental, untreated brain metastases that remain stable ≥ 4 weeks may participate in this study as long as they meet all of the following criteria:

   * No metastases to meninges, midbrain, pons, medulla oblongata, spinal cord or cerebellar metastases.
   * No compression of the aqueduct of Sylvius, no compression of the third or fourth ventricle, no compression of the spinal cord.
   * Total diameter of metastases ≤ 2 cm and total number of metastases ≤ 3.
   * After the completion of treatment for brain metastases, repeated imaging examination confirming no evidence of new brain metastases or enlargement of the original brain metastases must be ≥ 4 weeks from completion of radiotherapy (stereotactic radiosurgery or whole brain irradiation) using same imaging technique; no steroids, anticonvulsant, or dehydration (such as mannitol) therapy is required, and the symptoms are stable ≥ 14 days prior to randomization.
   * Measurable lesions per RECIST 1.1 excluding brain metastases.
4. Presence of any of the following hematologic abnormalities at Baseline*:

   * Hemoglobin < 9 g/dL.
   * Absolute neutrophil count (ANC) < 1,500 per mm3.
   * Platelet count <100 x 103/mm3. *""Baseline"" is defined as the last available observation prior to the first dose of investigational medical product. Note: Participants must not receive supportive treatments such as blood products (including red blood cell suspension, apheresis platelets, cryoprecipitation, etc.), erythropoietin, or colony-stimulating factors within 7 days prior to blood sampling.
5. Presence of any of the following serum chemistry abnormalities at Baseline:

   * Total bilirubin > 1.5 × upper limit of normal (ULN) except for participants with Gilbert's syndrome with serum bilirubin ≤ 3 × ULN or if concurrent conjugated bilirubin ≤ ULN.
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 × ULN; for liver metastasis, AST or ALT > 5.0 × ULN.
   * Creatinine Clearance (CrCl) < 30 mL/min; the Cockcroft-Gault formula is used to calculate CrCl (using ideal body weight for obese participants and actual body weight for non-obese participants).
   * Albumin < 30 g/L. Note: Investigators should refer to the local clinical practice guidelines or the label of docetaxel to assess whether participants with abnormal serum chemistry are suitable for docetaxel treatment.
6. Presence of any of the following coagulation parameter abnormalities at Baseline:

   * International normalized ratio (INR) > 1.5 × ULN (> 3 × ULN if on stable dose anticoagulation).
   * Partial thromboplastin time (PTT; or activated partial thromboplastin time [aPTT]) > 1.5 × ULN (> 3 × ULN if on stable-dose anticoagulation).
7. History of deep venous thrombosis, pulmonary embolism, or any other serious thromboembolic events within 3 months prior to enrollment (implantable port or catheter-related thrombosis, or superficial venous thrombosis are not considered ""serious"" thromboembolisms); portal vein tumor thrombus involving both the main trunk and bilateral first-order branches, or involving both the main trunk and superior mesenteric vein, or inferior vena cava tumor thrombus.
8. Active uncontrolled bleeding or known bleeding tendency. For example, imaging shows that the tumor invades large blood vessels or has unclear boundaries (including aorta, pulmonary aorta, left pulmonary artery, right pulmonary artery, pulmonary vein, superior vena cava, inferior vena cava, etc.), or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the subsequent study.
9. Presence of clinically significant cardiovascular or cerebrovascular diseases, including:

   * Symptomatic, clinically unstable arrhythmia or arrhythmia requiring clinical intervention.
   * Severe conduction disorders (such as third-degree atrioventricular block and bundle branch block).
   * QT interval corrected for heart rate (QTc interval, calculated using Fridericia's formula) ≥ 480 ms.
   * Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) despite standard treatment.
   * History of myocarditis.
   * Left ventricular ejection fraction (LVEF) < 50%.
   * Congestive heart failure requiring treatment.
   * Class II-IV cardiac insufficiency according to the New York Heart Association (NYHA) functional classification.
   * History of acute coronary syndrome (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to the first dose of investigational medical product.
   * Cerebrovascular accident or transient ischemic attack within 6 months before the first dose of the investigational medical product.
   * History of seizures.
10. Cardiac enzymes ≥ levels consistent with myocardial infarction as defined by the manufacturer (i.e., Grade 3).
11. History of the following lung diseases requiring steroid therapy: interstitial lung disease (ILD), pulmonary fibrosis, drug-related and radiation pneumonitis; current active pulmonary infection requiring anti-infective therapy; active pulmonary tuberculosis within 1 year prior to enrollment; severely impaired pulmonary function, including but not limited to the following: pulmonary embolism, severe asthma or chronic obstructive pulmonary disease within 3 months prior to randomization; autoimmune, connective tissue, or inflammatory diseases involving the lungs (such as rheumatoid arthritis, Sjögren's disease, and sarcoidosis); previous unilateral pneumonectomy.
12. History of severe, poorly controlled allergies, asthma or atopic dermatitis (except for atopic dermatitis caused by immunotherapy). Note: remote history of childhood asthma is not exclusionary.
13. History of anaphylactic or hypersensitivity reactions. Uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, abdominal effusion, pericardial effusion, etc.

    Note: Participants with the following conditions may be enrolled:
    * No need for drainage.
    * No significant increase in effusion after stopping drainage determined using at least 2 ultrasound examinations (at least 7 days apart).
14. Current or recent (within 6 months) significant gastrointestinal disease or condition, including:

    * Flare of inflammatory bowel disease.
    * Grade ≥ 2 diarrhea (CTCAE v5.0) within 2 weeks prior to the first dose of the investigational medical product.
15. Active autoimmune disease requiring systemic treatment (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose.

    Note: Replacement therapies (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments and exclusionary.
16. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
17. Known or suspected allergy to the investigational medical product and any excipients. Known or suspected severe hypersensitivity reactions to docetaxel or to drugs formulated with polysorbate 80.
18. Prior history of significant toxicity related to immune checkpoint inhibitor administration that required permanent discontinuation of this therapy.
19. Unresolved Grade > 1 toxicity related to any previous anti-tumor therapy (excluding alopecia, asthenia, hypothyroidism requiring only thyroid hormone replacement therapy, hyperglycemia requiring only insulin replacement therapy, adrenal insufficiency requiring physiological steroid replacement, electrolyte abnormalities requiring only symptomatic treatment, and other conditions not affecting the investigational medical product treatment as assessed by the investigator).
20. Have not adequately recovered from previous surgery or have undergone any major surgery, such as carotid artery stenting or esophageal stenting, within 4 weeks before the first dose of investigational medical product.
21. Uncontrolled tumor-related pain or symptomatic hypercalcemia.
22. Uncontrolled human immunodeficiency virus (HIV), active syphilis, active hepatitis B (HBV), hepatitis C (HCV), or tuberculosis.

    * Participants who are HIV-positive must have CD4 ≥ 350 cells/µL. Participants on established HAART (assuming no expected drug-drug interactions) for at least 4 weeks must an HIV viral load < 400 copies/mL.
    * Participants with positive results of Treponema pallidum haemagglutination (TPHA)/Treponema pallidum particle agglutination (TPPA) test and/or rapid plasma regain test (RPR) should not be enrolled.
    * Participants with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) should undergo hepatitis B virus (HBV) DNA testing. If the HBV DNA copy number is ≤ 2.5 × 103 copies/mL or ≤ 500 IU/mL or below the lower limit of detection, the participant can be enrolled. Participants who are HBsAg (+) should receive anti-HBV treatment throughout the Treatment Period to avoid viral activation. For participants with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV treatment can be considered but is not required; however, close monitoring for viral reactivation is required.
    * Participants with positive HCV serology results but negative or below the lower limit of detection of HCV RNA can be included in the study.
    * Participants who received HCV treatment and have undetectable viral load results are allowed.
    * Participants with previously cured or clinically stable remote history of tuberculosis as assessed by the investigator can be included in the study.
23. Serious/active/uncontrolled infection, infection requiring systemic intravenous antibiotics, or fever of unknown origin (≥ 38°C) within 2 weeks before the first dose of investigational medical product(s).
24. History or current evidence of any disease, treatment, or laboratory abnormality that, in the judgment of the investigator, could compromise the safety of the participant, interfere with obtaining informed consent, affect participant compliance, or affect safety evaluations of the investigational medical product.
25. Psychiatric illness, altered mental status, or drug abuse that prevents understanding of the informed consent process and/or completion of required study-related evaluations.
26. Unable to meet protocol requirements for known or foreseeable reasons per investigator judgement.
27. Diagnosed with other pathologically confirmed malignancies within 5 years prior to informed consent, with the exception of radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ, localized prostate cancer, papillary thyroid cancer, and other radically treated malignancies with no known active disease for at least 2 years prior to enrollment and with a very low risk of recurrence.
28. Received any of the following excluded medications or treatments:

    * Docetaxel.
    * Received more than one anti-PD-1/PD-L1 monoclonal antibody therapy.
    * Systemic anti-tumor therapy except anti-PD-1/PD-L1 monoclonal antibody and platinum-based doublet chemotherapy including but not limited to bispecific antibodies, targeted therapy, antibody drug conjugate, other immune checkpoint inhibitors.
    * IL-2/IL-15 cytokine.
    * Chemotherapy within 2 weeks or 5 half-lives (whichever is longer) before the first dose of investigational medical product without delayed toxicity.
    * Anti-tumor antibody therapy (excluding antibody drugs such as denosumab for the treatment of bone metastases) within 4 weeks before the first dose of the investigational medical product.
    * Palliative radiotherapy within 2 weeks prior to the first dose of investigational medical product.
    * Live vaccine within 28 days prior to the first dose of investigational medical product.
    * Immunosuppressive or systemic steroid therapy (> 10 mg/day of prednisone or equivalent) within 2 weeks prior to the first dose of investigational medical product.
    * Received traditional Chinese medicine with anti-tumor indications within 1 week before the first dose of the investigational medical product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 37 Months from First Patient In (FPI) (event driven)
  To compare the overall survival (OS) of IBI363 (treatment group) vs. docetaxel (control group) in participants with unresectable locally advanced or metastatic squamous NSCLC with disease progression on or after platinum-based chemotherapy and anti-PD-1/PD-L1 immunotherapy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 44 months
  investigator assessed PFS per RECIST v1.1
Objective Response Rate (ORR) | 44 months
  the proportion of participants with a best overall response of complete response (CR) or partial response (PR), per RECIST v1.1.
Disease Control Rate (DCR) | 44 months
  the proportion of participants who achieve CR, PR, or stable disease (SD), per RECIST v1.1.
Duration of Response (DOR) | 44 momths
  time of first documented CR or PR to the time of disease progression or death
Time to Response (TTR) | 44 months
  time from randomization to the first occurrence of a response (CR or PR), per RECIST v1.1.
Safety Profile | 44 months
  percentrage of participants with: TEAEs/TRAEs any grade / ≥ grade 3; TESAEs/TRSAEs; AESI (adverse events of special interest as defined in protocol); irAEs any grade/ ≥ gr 3; TEAEs/TRAEs leading to interruption/discontinuation/death; infusion related reactions any grade/ ≥ grade 3
Pharmacokinetic parameters including Terminal Half-Life (t½) of IBI363 | 44 months
  The terminal elimination half-life will be calculated from the terminal phase of the plasma concentration-time curve.
Pharmacokinetic parameters including Clearance (CL) of IBI363 | 44 months
  Clearance will be calculated using dose/AUC.
Pharmacokinetic parameters including Volume of Distribution (Vd) of IBI363 | 44 months
  Volume of distribution will be estimated based on non-compartmental analysis.
Number of Participants Who Develop Anti-Drug Antibodies (ADA) to IBI363 (immunogenicity) | 44 months
  Positive rates of anti-IBI363 antibody (ADA) and/or neutralizing antibody (NAb) in participants receiving IBI363 are planned to evaluate.
Change from Baseline in Global Health Status / Quality of Life (QoL) Score Using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 44 months
  Global Health Status / Quality of Life (QoL) will be assessed using the EORTC QLQ-C30. Scores range from 0 to 100. For the Global Health Status/QoL scale, a higher score indicates a better outcome (i.e., better QoL). The change from baseline to each time point will be analyzed.

OTHER OUTCOMES:
Exploratory: Baseline and Time to Deterioration in EORTC QLQ-C30 Global Health Status / Quality of Life (QoL) Score | 44 months
  Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores range 0-100; higher scores indicate better QoL. Time to deterioration is defined as the time from baseline to a clinically meaningful decline in score.
Exploratory: Baseline and Time to Deterioration in EORTC QLQ-C30 Symptom and Functional Scales | 44 monthd
  Patient-reported symptoms (e.g., fatigue, pain) and functioning (e.g., physical, emotional) will be assessed using subscales of the EORTC QLQ-C30. Scores range 0-100; higher symptom scores indicate worse symptoms, higher functioning scores indicate better functioning. Time to deterioration defined as time to clinically meaningful decline.
Exploratory: Baseline and Time to Deterioration in EQ-5D-5L Index Score | 44 months
  Health-related quality of life will be assessed using the EuroQoL-5-Dimensions 5-Level questionnaire (EQ-5D-5L). The index score ranges from -0.594 to 1, where 1 indicates perfect health. Time to deterioration is defined as the time to a clinically meaningful decrease in the index score.
Exploratory: Baseline and Time to Deterioration in EQ-5D-5L Visual Analog Scale (VAS) Score | 44 months
  The EQ-5D-5L includes a Visual Analog Scale (VAS) where participants rate their overall health from 0 (worst) to 100 (best). Time to deterioration defined as time to meaningful decrease in VAS score.
Exploratory: Correlation Between PD-L1 Expression in Tumor Tissue and Objective Response Rate (ORR) to IBI363 | 44 months
  PD-L1 expression will be measured by immunohistochemistry (IHC) using [specify assay if known, e.g., 22C3 pharmDx]. Expression will be correlated with objective response rate (ORR) per RECIST v1.1.
Exploratory: Correlation Between Baseline Immune Cell Infiltration and Progression-Free Survival (PFS) in Participants Treated with IBI363 | 44 momths
  PD-L1 expression will be measured by immunohistochemistry (IHC) using 22C3 pharmDx. Expression will be correlated with progression-free survival (PFS) assessed per RECIST v1.1.
Exploratory: Correlation Between PD-L1 Expression and Incidence of Treatment-Emergent Adverse Events (TEAEs) | 44 months
  PD-L1 expression (via IHC) will be correlated with the incidence of treatment-emergent adverse events (TEAEs), graded per CTCAE v5.0.
Exploratory: Correlation Between Baseline Immune Cell Infiltration and Objective Response Rate (ORR) to IBI363 | 44 months
  Immune cell infiltration (e.g., CD8+ T cells, CD4+ T cells) will be quantified by immunohistochemistry (IHC) or multiplex immunofluorescence (mIF). Results will be correlated with objective response rate (ORR) assessed per RECIST v1.1.
Exploratory: Change from Baseline in Serum Cytokine Levels Following IBI363 Administration | 44 months
  Cytokine concentrations will be measured in serum using a validated multiplex immunoassay. Changes from baseline will be used to assess pharmacodynamic effects of IBI363.
Exploratory: Change from Baseline in Soluble CD25 (sCD25) Levels in Peripheral Blood Following IBI363 Administration | 44 months
  Soluble CD25 (sCD25) concentrations will be measured in serum using a validated immunoassay. Changes from baseline will be analyzed as a pharmacodynamic biomarker of IL-2 pathway activation.
Exploratory: Change from Baseline in RNA Expression Profiles of Peripheral Immune Cells Following IBI363 Treatment | 44 months
  RNA from peripheral blood mononuclear cells (PBMCs) will be isolated and analyzed using bulk RNA sequencing. Differential gene expression and pathway enrichment analyses will be performed to evaluate pharmacodynamic effects of IBI363.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Memorial Health Services, Fountain Valley, California
  - BRCR Global, Tamarac, Florida
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China